CLINICAL TRIAL: NCT02758626
Title: A Phase 2 Randomized, Double-Masked Placebo-Controlled Crossover Safety and Tolerability Study of Ataluren for Drug Resistant Epilepsy in Patients With Nonsense Mutation CDKL5 or Dravet Syndrome
Brief Title: Ataluren for Nonsense Mutation in CDKL5 and Dravet Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-00426
Record Dates: First submitted 2016-04-04; First posted 2016-05-02 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — ataluren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ataluren Followed By Placebo (Active Comparator): Cross Over Design: Treatment Period 1 with Ataluren (Week 0/Day 1 to Week 12), Washout Period (Week 12 to Week 16), crossover to Placebo Treatment Period 2 (Week 16 to Week 28), and Follow-up (Week 28 to Week 32).
  Interventions: Drug: ataluren; Drug: Placebo
- Placebo Followed by Ataluren (Active Comparator): Treatment Period 1 with Placebo (Week 0/Day 1 to Week 12), Washout Period (Week 12 to Week 16), crossover to Treatment Period 2 with Ataluren(Week 16 to Week 28).
  Interventions: Drug: ataluren; Drug: Placebo

INTERVENTIONS:
Drug: ataluren — Powder formulation
  Other Names: PTC124
Drug: Placebo — Powder formulation

SUMMARY:
This is a phase 2, crossover study of Ataluren for the treatment of nonsense mutation Dravet syndrome or cyclin-dependent kinase-like 5 (CDKL5) deficiency, resulting in drug-resistant epilepsy. Patients will receive 12 weeks of ataluren or placebo during each treatment period. Treatment Period 1 will be followed by a 4-week Washout Period. Based on ataluren PK and pharmacodynamic data, the 4-week washout period is deemed an appropriate length of time to eliminate any ataluren drug effects. Following the Washout Period, patients will crossover to receive the opposite treatment during Treatment Period 2 as follows: Patients receiving ataluren during Treatment Period 1 will receive placebo during Treatment Period 2. Patients receiving placebo during Treatment Period 1 will receive ataluren during Treatment Period 2.

DETAILED DESCRIPTION:
Investigators will try to characterize the safety profile of ataluren in patients with CDKL5 or Dravet syndrome resulting from a nonsense mutation and evaluate changes in convulsive and/or drop seizure frequency from Baseline following ataluren treatment in patients with CDKL5 or Dravet syndrome resulting from a nonsense mutation. Investigators will measure changes in minor seizure types (absence, myoclonic, complex partial/focal dyscognitive) following ataluren treatment in patients with CDKL5 or Dravet syndrome resulting from a nonsense mutation and changes from Baseline in cognitive, motor, and behavioral function as well as QOL following ataluren treatment in patients with CDKL5 or Dravet syndrome resulting from a nonsense mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 years old and ≤ 12 years old, male or female, at Week 0 (at time informed consent/assent is signed)
2. Documentation of a diagnosis of Dravet syndrome or CDKL5 deficiency resulting from a nonsense mutation in 1 allele, as evidenced by medical records, genetic testing, and the following clinical feature:

   a. Failure to control seizures despite appropriate trial of 2 or more AEDs at therapeutic doses
3. Between 1 to 3 baseline AEDs at stable doses for a minimum for 4 weeks prior to the Baseline visit

   a. Vagus nerve stimulator (VNS), ketogenic diet, and modified Atkins diet do not count towards this limit but must be unchanged for 3 months prior to enrollment (Baseline).
4. VNS must be on stable settings for a minimum of 3 months prior to the Baseline visit
5. If on ketogenic or modified Atkins diet, must be on stable ratio for a minimum of 3 months prior to the Baseline visit
6. Written consent obtained from the patient or patient's legal representative must be obtained prior to performing any study procedures
7. Minimum of 6 convulsive or drop seizures with duration > 3 seconds over the 4 weeks of diary screening prior to randomization and ≥ 6 convulsive or drop seizures with duration > 3 seconds during the 4 weeks from Screening to Baseline.

Exclusion Criteria:

1. Patient is < 2 years old or ≥ 12 years old
2. Epilepsies associated with genetic disorders other than Dravet syndrome or CDKL5 deficiency
3. Patient has Dravet or CDKL5 genetic mutations that are NOT nonsense mutations
4. Felbatol has been initiated within the past 12 months prior to the Screening Visit
5. Patients who are currently or have participated in clinical trials in the 30 days prior to enrollment (Baseline Visit)
6. Prior or ongoing medical condition (eg, concomitant illness, psychiatric condition), medical history, physical findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the patient, makes it unlikely that the course of study drug administration or follow-up would be completed, or could impair the assessment of study results.
7. Ongoing intravenous administration of aminoglycosides or vancomycin.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-11; Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orrin Devinsky, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Devinsky O, King L, Bluvstein J, Friedman D. Ataluren for drug-resistant epilepsy in nonsense variant-mediated Dravet syndrome and CDKL5 deficiency disorder. Ann Clin Transl Neurol. 2021 Mar;8(3):639-644. doi: 10.1002/acn3.51306. Epub 2021 Feb 4. PMID 33538404

RESULTS

PARTICIPANT FLOW:
Groups:
- Ataluren Followed By Placebo: Cross Over Design: Treatment Period 1 with Ataluren (Week 0/Day 1 to Week 12), Washout Period (Week 12 to Week 16), crossover to Placebo Treatment Period 2 (Week 16 to Week 28), and Follow-up (Week 28 to Week 32). Participants have option to enroll in open-label extension (OLE) at Week 28. During the OLE, all participants receive open-label Ataluren.
  ataluren: Powder formulation. Dose: 3 times per day (TID; 10 mg/kg, 10 mg/kg, and 20 mg/kg at morning, midday, and evening, respectively)
  Placebo: Powder formulation. Dose: 3 times per day (TID; 10 mg/kg, 10 mg/kg, and 20 mg/kg morning, midday, and evening, respectively)
- Placebo Followed by Ataluren: Cross Over Design: Treatment Period 1 with Placebo (Week 0/Day 1 to Week 12), Washout Period (Week 12 to Week 16), crossover to Treatment Period 2 with Ataluren(Week 16 to Week 28). Participants have option to enroll in open-label extension (OLE) at Week 28. During the OLE, all participants receive open-label Ataluren.
  ataluren: Powder formulation. Dose: 3 times per day (TID; 10 mg/kg, 10 mg/kg, and 20 mg/kg at morning, midday, and evening, respectively)
  Placebo: Powder formulation. Dose: 3 times per day (TID; 10 mg/kg, 10 mg/kg, and 20 mg/kg morning, midday, and evening, respectively)
Period: Double-Blind Phase (Week 0 - Week 28)
Arm/Group | Ataluren Followed By Placebo | Placebo Followed by Ataluren
Started | 9 | 6
Completed | 8 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Open-Label Extension (Week 28-Week 124)
Arm/Group | Ataluren Followed By Placebo | Placebo Followed by Ataluren
Started | 8 | 6
Completed | 6 | 3
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Parental/Legal Guardian withdrawal of consent | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ataluren Followed By Placebo | Placebo Followed by Ataluren | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (4.7) | 12.0 (0.0) | 10.4 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in 28-Day Convulsive Seizure Frequency During Ataluren Treatment Period
Description: Convulsive seizure frequency per 28 days is defined as total number of convulsive seizures reported during the period divided by number of days during the period seizures were assessed, multiplied by 28. Percent change from Baseline will be defined as the frequency of seizures per 28 days during the Ataluren Treatment Period minus frequency of seizures per 28 days at Baseline, divided by the frequency of seizures per 28 days at Baseline, multiplied by 100. Negative percent change from Baseline indicates improvement.
Time Frame: Baseline, Week 12 of Ataluren Treatment (Up to Week 28)
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Ataluren: 12-week treatment regimen.
Arm/Group | Ataluren
Number analyzed (Participants) | 14
percent change | 723.17 (279.912)

2. Primary Outcome: Percent Change From Baseline in 28-Day Convulsive Seizure Frequency During Placebo Treatment Period
Description: Convulsive seizure frequency per 28 days is defined as total number of convulsive seizures reported during the period divided by number of days during the period seizures were assessed, multiplied by 28. Percent change from Baseline will be defined as the frequency of seizures per 28 days during the Placebo Treatment Period minus frequency of seizures per 28 days at Baseline, divided by the frequency of seizures per 28 days at Baseline, multiplied by 100. Negative percent change from Baseline indicates improvement.
Time Frame: Baseline, Week 12 of Placebo Treatment (Up to Week 28)
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo: 12-week treatment regimen.
Arm/Group | Placebo
Number analyzed (Participants) | 14
percent change | 0.72 (222.82)

ADVERSE EVENTS:
Time Frame: up to Year 1
Arm/Group | Ataluren | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 7/15 | 1/14
Other Adverse Events (participants affected / at risk) | 13/15 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=15) | Placebo (N=14)
Influenza (Infections and infestations) | 2 | 1
Croup Infections (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Pneumonia Mycoplasmal (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Drug Level Decreased (Investigations) | 3 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Seizures (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=15) | Placebo (N=14)
Viral upper respiratory tract infection (Infections and infestations) | 9 | 2
Camphylobacter gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteriritis viral (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 5 | 2
Viral infection (Infections and infestations) | 1 | 1
Croup infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Pnuemonia mycoplasmal (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 4
Flatulence (Gastrointestinal disorders) | 4 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Eructation (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Gastroesophagael reflux disease (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 12 | 2
Fatigue (General disorders) | 1 | 1
Increased Drug level (Investigations) | 2 | 0
Body temperature increased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Increased seizures (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 4 | 0
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0
Drooling (Nervous system disorders) | 1 | 1
Seizures (Nervous system disorders) | 5 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Tics (Psychiatric disorders) | 1 | 0
Screaming (Psychiatric disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Pollakuria (Renal and urinary disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin warm to touch (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Multiple allergies (Immune system disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT02758626/Prot_SAP_000.pdf